CLINICAL TRIAL: NCT00505258
Title: Randomized, Open-Label Study Evaluating the Safety and Rate of Bacterial Clearance of Ceftobiprole 500 Milligram Every 8 Hours Compared to Conventional Therapy in the Treatment of Hospitalized Subjects With Staphylococcus Aureus Bacteremia
Brief Title: Ceftobiprole in the Treatment of Hospitalized Patients With Staphylococcus Aureus Bacteremia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was withdrawn due to lack of an appropriate patient population.
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR013807
Record Dates: First submitted 2007-07-19; First posted 2007-07-23 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Bacteremia
Keywords: Bacteremia; Bloodstream infection; Staphylococcus aureus; Staphylococcal Infections; MRSA; MSSA
MeSH Terms: conditions — Bacteremia; Sepsis; Staphylococcal Infections | interventions — ceftobiprole medocaril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ceftobiprole medocaril

SUMMARY:
The purpose of this study is to assess the safety and efficacy of ceftobiprole versus a comparator in hospitalized patients with bacteremia.

DETAILED DESCRIPTION:
Ceftobiprole medocaril is a cephalosporin antibiotic with anti-MRSA (Methicillin-Resistant Staphylococcus aureus) activity. Ceftobiprole medocaril in not approved for the treatment of bacterial blood stream infections. S. aureus is a major human pathogen. It causes a wide range of serious infections, including skin and skin structure infections, infections of vascular devices and catheters, and infections of the heart and lungs, bones and joints, and deep tissues. Particularly challenging and difficult to treat are blood-borne infections (bacteremia). Bacteremic infections are prone to relapse and they are often complicated by metastatic seeding of sites throughout the body. MRSA strains are increasing in prevalence, incidence, and virulence. Moreover, the frequency of patients presenting with persistent MRSA bacteremia appears to be rising. The objective of the open label trial is to compare the effectiveness and safety of ceftobiprole versus a comparator in patients with MRSA and MSSA (methicillin-susceptible Staphylococcus aureus) in bacteremic patients. Patients who meet inclusion and exclusion criteria and consent to participate in the study will be randomly assigned to either ceftobiprole or comparator. The primary end point is time to bloodstream clearance of MRSA and MSSA in patients. Patients will be randomized to either ceftobiprole or comparator for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with signs and symptoms suggestive of systemic staphylococcal infection as defined in the protocol
* Female patients must be postmenopausal (for at least 1 year), surgically sterile or practicing an effective method of birth control, male partner sterilization or, at the discretion of the investigator, abstinence, before entry and throughout the study and have a negative urine pregnancy test (confirmed with a negative serum pregnancy test) at screening.

Exclusion Criteria:

* Female patients who are pregnant or lactating
* Known or suspected hypersensitivity to beta-lactam antibiotics or any other study medications
* Receipt of vancomycin or other antistaphylococcal drug for > 2 calendar days prior to initiation of study drug
* Diagnosis of a catheter-related GPC-cl bacteremia at the time of study enrollment
* Clinical findings of left-sided endocarditis prior to enrollment or any time during study participation
* Requirement for surgery during the seven days of study therapy administration with the exception of surgery required to manage a complication of S. aureus bacteremia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
To determine the effect of ceftobiprole on the time to bloodstream clearance of methicillin-resistant Staphylococcus aureus and methicillin-susceptible Staphylococcus aureus (MSSA) in treated bacteremic patients.

SECONDARY OUTCOMES:
To determine the effect of ceftobiprole versus comparator on the time to bloodstream clearance of MRSA and MSSA, respectively and bloodstream clearance of MRSA compared to MSSA in bacteremic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ortho-McNeil Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Ortho-McNeil Janssen Scientific Affairs, LLC